CLINICAL TRIAL: NCT02519049
Title: Diagnostic and Prognostic Role of 11C-Methionine PET/CT Imaging in Patients Affected by Malignant Pleural Mesothelioma (MPM) and Candidate to Pleurodesis
Brief Title: 11C-Methionine PET/CT Imaging in Patients Affected by Malignant Pleural Mesothelioma (MPM)
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 1287
Record Dates: First submitted 2015-06-26; First posted 2015-08-10 (Estimated); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Mesothelioma, Malignant
Keywords: Mesothelioma; 11C-methionine PET; talc pleurodesis
MeSH Terms: conditions — Mesothelioma, Malignant; Mesothelioma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biopsy specimen
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention — This is an observational study

SUMMARY:
Prospective exploratory study specifically investigating the role of 11C-Methionine PET/CT imaging in patients affected by Malignant Pleural Mesothelioma (MPM) and candidate to pleurodesis.

DETAILED DESCRIPTION:
This is a single-center, open-label study, lasting 36 months including an estimated period of 24 months for the enrollment and max 12 months of follow-up. All patients affected by MPM and referred to our Institution eligible for therapeutic pleurodesis and subsequent platinum- and pemetrexed-based chemotherapy will be enrolled. In all cases patients will be investigated with 11C-Methionine PET/CT and 18F-FDG PET/CT before talc pleurodesis, one week after and at the end of three cycles of chemotherapy.

A minimum number of 20 patients will be considered for the analysis.

ELIGIBILITY:
Inclusion Criteria:

* patients with an histological diagnosis of MPM eligible for pleurodesis and scheduled to undergo platinum- and pemetrexed-based chemotherapy.
* obtained informed consent

Exclusion Criteria:

* patients age <18 years
* pregnancy or breast-feeding;
* patients affected by other malignancies within the last 3 years;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients affected by MPM and referred to our Institution for therapeutic pleurodesis and subsequent platinum- and pemetrexed-based chemotherapy will be enrolled. A minimum number of 20 patients will be considered for the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-09; Primary Completion 2018-09 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Variation of SUVmax (Maximal Standardized Uptake Value) in patients undergoing talc pleurodesis | Change from Baseline in SUVmax up to 1 week after talc pleurodesis.

CONTACTS AND LOCATIONS:
Overall Officials: Egesta Lopci, MD, Principal Investigator — Humanitas Clinical and Research Hospital
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

REFERENCES:
- [Background] Lopci E, Zucali PA, Ceresoli GL, Perrino M, Giordano L, Gianoncelli L, Lorenzi E, Gemelli M, Santoro A, Chiti A. Quantitative analyses at baseline and interim PET evaluation for response assessment and outcome definition in patients with malignant pleural mesothelioma. Eur J Nucl Med Mol Imaging. 2015 Apr;42(5):667-75. doi: 10.1007/s00259-014-2960-y. Epub 2014 Nov 18. PMID 25403555
- [Background] Ceresoli GL, Chiti A, Zucali PA, Cappuzzo F, De Vincenzo F, Cavina R, Rodari M, Poretti D, Lutman FR, Santoro A. Assessment of tumor response in malignant pleural mesothelioma. Cancer Treat Rev. 2007 Oct;33(6):533-41. doi: 10.1016/j.ctrv.2007.07.012. Epub 2007 Aug 30. PMID 17764849
- [Background] Ceresoli GL, Chiti A, Santoro A. 11C-labeled methionine and evaluation of malignant pleural mesothelioma. N Engl J Med. 2007 Nov 8;357(19):1982-4. doi: 10.1056/NEJMc071823. No abstract available. PMID 17989397
- [Background] Lopci E, Novellis P, Testori A, Rahal D, Voulaz E, Bottoni E, Ferraroli GM, Crepaldi A, Ceresoli GL, Perrino M, Castello A, Alloisio M, Veronesi G, Zucali PA. In-vivo imaging of methionine metabolism in patients with suspected malignant pleural mesothelioma. Nucl Med Commun. 2019 Nov;40(11):1179-1186. doi: 10.1097/MNM.0000000000001078. PMID 31568271
- [Background] Zucali PA, Lopci E, Ceresoli GL, Giordano L, Perrino M, Ciocia G, Gianoncelli L, Lorenzi E, Simonelli M, De Vincenzo F, Setti LR, Bonifacio C, Bonomi M, Bombardieri E, Chiti A, Santoro A. Prognostic and predictive role of [18 F]fluorodeoxyglucose positron emission tomography (FDG-PET) in patients with unresectable malignant pleural mesothelioma (MPM) treated with up-front pemetrexed-based chemotherapy. Cancer Med. 2017 Oct;6(10):2287-2296. doi: 10.1002/cam4.1182. Epub 2017 Sep 21. PMID 28941158
- [Background] Bonomi M, De Filippis C, Lopci E, Gianoncelli L, Rizzardi G, Cerchiaro E, Bortolotti L, Zanello A, Ceresoli GL. Clinical staging of malignant pleural mesothelioma: current perspectives. Lung Cancer (Auckl). 2017 Aug 18;8:127-139. doi: 10.2147/LCTT.S102113. eCollection 2017. PMID 28860886